CLINICAL TRIAL: NCT02793258
Title: Impact of Transcranial Direct Current Stimulation on Emotional Processing in Major Depression
Brief Title: Impact of tDCS on Emotional Processing in Major Depression
Acronym: EmoStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-A00415-46
Record Dates: First submitted 2016-05-18; First posted 2016-06-08 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Major Depressive Disorder
Keywords: tDCS; neuromodulation; depression; cognition
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo tDCS (Placebo Comparator): Subjects will receive 10 30-minutes sessions of sham tDCS, twice a day for 5 consecutive day.
  Facial emotion recognition task and attentional task with measurement of eye-tracking, heartrate, respiratory frequency and skin conductance will be conducted before and after the first session, and after the last session.
  Interventions: Device: transcranial direct current stimulation
- Active tDCS (Experimental): receive 10 30-minutes sessions of two milliamps tDCS, twice a day for 5 consecutive day.
  Stimulation will be performed using an tDCS stimulator with two 7×5 cm (35 cm2) sponge electrodes soaked in a saline solution (0.9% NaCl) Anode will be placed over the left dorsolateral prefrontal cortex (F3 according to the international EEG system) and cathode over the right dorsolateral prefrontal cortex (F4 according to the international EEG system) The twice daily sessions will be separated by at least 2 hours.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Subjects will receive 10 30-minutes sessions of two milliamps transcranial direct current stimulation , twice a day for 5 consecutive day.
  Facial emotion recognition task and attentional task with measurement of eye-tracking, heartrate, respiratory frequency and skin conductance will be conducted before and after the first session, and after the last session.

SUMMARY:
Background: transcranial direct current stimulation (tDCS) is an innovative treatment for major depression. However, its mechanisms of action are still unclear. Major depression is characterized by impaired processing of emotional information, which returns back to normal after successful antidepressant treatment. In this randomized double-blind study, the investigators aim to assess the effect of tDCS on emotional processing in major depression.

DETAILED DESCRIPTION:
Methods: 40 subjects with major depression (20 active treatment and 20 placebo) will receive ten 30-minutes sessions of active two milliamps or sham tDCS (anode over left dorsolateral prefrontal cortex and cathode over right dorsolateral prefrontal cortex), twice a day for 5 consecutive days. Psychometric assessment of depression (MADRS,Beck Depression Inventory , CGI) and a neuropsychological assessment will be conducted before and after the treatment.

A facial emotion recognition task and an attentional emotional task with measurement of eye-tracking, heart rate, respiratory frequency and skin conductance will be conducted before and after the first session, and after the last session.

The investigators hypothesize that active tDCS will improve emotional processing in major depression, and that this will be observed after 1 and 10 sessions of tDCS.

Conclusions: Studying the impact of transcranial direct current stimulation on emotional processing in major depression could allow to better understand its antidepressant mechanisms

ELIGIBILITY:
Inclusion Criteria:

Healthy controls:

* Age between 18 and 65 years
* Given consent.

Depressed subjects:

* Major depressive episode (no psychotic features) according to Diagnostic ans Statistical of Mental Disorders number 5 (DSM 5.0.)
* Age from 18-65
* Antidepressant stable for the last 4 weeks
* MADRS ≥ 20.
* Given consent

Exclusion Criteria:

Healthy controls:

* Psychiatric disorder
* Addiction except for tobacco addiction
* Ocular disease (except from refraction disorders), neurologic or cardiac disease.
* Neuroleptic or anticonvulsivant treatment
* Presence of a specific contraindication for tDCS (e.g., personal history of epilepsy, metallic head implant, cardiac pacemaker)

Depressed subjects:

* Other psychiatric disorder except for personality disorders
* Ocular disease (except from refraction disorders), neurologic or cardiac disease.
* Neuroleptic or anticonvulsivant treatment
* Presence of a specific contraindication for tDCS (e.g., personal history of epilepsy, metallic head implant, cardiac pacemaker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Number of correct responses at a facial expression recognition task | within 5 days after stimulation
  A computerized facial expression recognition task was designed for the study. 240 pictures of emotional faces (8 identities, expressing anger, sadness, happiness, surprise, disgust, or fear, morphed with intensity of 20, 40, 50, 60 and 80%) are randomly displayed on a screen for 500ms. Subjects are asked to identify the emotion by answering on a keyboard.
  Rate of correct responses is the main outcome. During this task, eye movements are recorded by an eye-tracking device. Skin conductance, respiratory and heart rate frequency are also recorded

SECONDARY OUTCOMES:
Evolution of the depressive symptoms measured by MADRS | an average of two weeks
  Montgomery-Asberg Depression Rating Scale is a 10-item scale to evaluate the intensity of the depressive symptoms.
Performance on an attentional dot-probe task | within 5 days after stimulation
  Computerized "dot-probe " attentional task designed for the study. Pairs of emotional faces (neutral/sad ou neutral/happy) are randomly presented on a screen for 1000ms. Then, a probe is presented during 1100ms.subjects are asked to indicate a which side the probe approved During this task, eye movements are recorded by an eye-tracking device. Total time spent on Region of Interest (sad, happy or neutral face) is measured.
  Skin conductance, respiratory and heart rate frequency are also recorded.
tests of executive functions | an average of two weeks
  Neuropsychological assessment : attentional functioning (TAP), executive functioning (BADS, working memory, go/no-go, stroop), memory (california verbal learning test) Improvement of executive functioning by tDCS will be assessed.
Beck depression inventory scale | within 5 days after stimulation
Clinical global impression scale | an average of two weeks
Eye movements during facial emotion recognition task and attentional task | within 5 days after stimulation
  Recorded by Eye tracker.Measurement of total time spent on specific Region of interest (eyes, nose, mouth, emotional face)
Skin conductance measured in speed per microseconds | within 5 days after stimulation
  Recorded with physiologic data system (BIOPAC)
Heart rate measured in number of heart pulses per milliseconds | within 5 days after stimulation
  Recorded with physiologic data system (BIOPAC)
Respiratory frequency measured in number of respiratory cycles per minute | within 5 days after stimulation
  Recorded with physiologic data system(BIOPAC)

CONTACTS AND LOCATIONS:
Overall Officials: HAESEBAERT FREDERIC, PH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Ch Le Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Equip (PSYR2) -Psychiatric Disorders: from Resistance to Response — http://www.ch-le-vinatier.fr/offre-de-soins/la-recherche/les-equipes/equipe-psr2-706.html